CLINICAL TRIAL: NCT06492421
Title: Phase II Study of Neoadjuvant CT-Guided Intra-tumor Double Checkpoint Blockades for Untreated Stage I-IIIA Non-Small Cell Lung Cancers Amenable for Surgical Resection
Brief Title: Neoadjuvant Intra-tumor Double Immunotherapy for Lung Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZ-IT-ICIs-LC-Neoadjuvant-028
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Surgery; Non-small Cell Lung Cancer
Keywords: NSCLC; Intra-tumor injection; Neoadjuvant therapy; Double immunotherapy; Interventional radiology; Bevacizumab
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; pembrolizumab; durvalumab; Idarubicin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: IT injection of double ICIs (Experimental): Neoadjuvant therapy: intra-tumor injection of double ICIs only.
  Interventions: Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab
- Group 2: IT injection of double ICIs and chemodrug (Experimental): Neoadjuvant therapy: intra-tumor injection of double ICIs and chemodrug.
  Interventions: Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab
- Group 3: IT injection of double ICIs and chemodrug plus bevacizumab (Experimental): Neoadjuvant therapy: intra-tumor injection of double ICIs and chemodrug plus bevacizumab.
  Interventions: Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab

INTERVENTIONS:
Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab — This study has 3 subgroups:
  Arm 1. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab is administrated with a total dose of 1-2mg/kg via intra-tumor fine needle injection in 10 min, every 3 weeks, total 3-4 times.
  Arm 2. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab combined with idarubicin is administrated via intra-tumor fine needle injection in 15 min, every 3 weeks, total 3-4 times.
  Arm 3. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab combined with idarubicin plus bevacizumab is administrated via intra-tumor fine needle injection in 20 min, every 3 weeks, total 3-4 times.
  Other Names: Other ICIs

SUMMARY:
This phase II trial studies how well intra-tumor injection of double checkpoint inhibitors work when given alone and in combination with chemotherapy or/and bevacizumab in treating patients with previously untreated stage I-IIIA non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as ipilimumab, pembrolizumab or durvalumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Drugs used in interventional radiological chemotherapy, such as idabubicin, can directly kill the cancer cell and release tumor antigens to activate DC function in situ. Giving intra-tumor injection of checkpoints inhibitors with or without chemotherapy and/or bevecizumab may work better than in vein infusion of the drugs in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Antibodies against CTLA4, PD1 or PDL1 are representative drugs for the check-points inhibitory agents, and their clinical indications have been approved in various types of tumors, including advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients, et al. Those drugs are regularly systemically administrated by vein infusion, however, local delivery of those drugs via interventional radiology technique including trans-artery or intra-tumor injection may increase the local drug concentration of the tumor, improve the efficacy, and reduce systemic adverse reactions. CTLA4 antibody ipilimumab has been widely effectively using to combine with PD1 or PDL1 antibody and this study is to combine ipilimumab and PD1 antibody or PDL1 antibody, so called double checkpoint inhibitors combination therapy, as neoadjuvant therapy for NSCLC via intra-tumor admistration. To the investigator's knowledge, no studies have been developed on the safety, efficacy and survival benefit of the double checkpoint inhibitors combination therapy for cancer patients as neoadjuvant treatment via intra-tumor delivery. This phase II clinical trial is designed to assess the safety and survival benefit of ipilimumab and pembrolizumab or durvalumab combination with or without chemodrug and/or bevacizumab as neoaduvant therapy on patients with NSCLC, including safety, pCR, mPR, PFS, ORR, DCR, and median survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed previously untreated non-small cell lung cancer. If a diagnostic biopsy is available, a pre-treatment biopsy is not required. Patients with a suspected lung cancer are eligible, but pathology must be confirmed prior to initiating treatment on study.
2. Patients with stage IIIA must not have more than one mediastinal lymph node station involved by tumor.
3. All patients must have lymph node evaluation of contralateral stations 2 and/or 4 to exclude N3 disease.
4. The patient must be a suitable candidate for surgery, in the opinion of the treating physician.
5. Signed and dated written informed consent must be provided by the patient prior to admission to the study in accordance with International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines and to the local legislation.
6. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1.
7. Absolute neutrophil count (ANC) >= 1.5 x 10^9/L; Hemoglobin >= 8.0 g/dL; Platelets >= 100 x 10^9/L; Total bilirubin =< 1.5 x upper limit of normal (ULN) (except subjects with Gilbert syndrome who can have total bilirubin < 3.0 mg/dL); Creatinine =< 1.5 x ULN or calculated creatinine clearance >= 50 mL/min using Cockcroft-Gault formula for creatinine clearance calculation OR 24-hour urine creatinine clearance >= 50 mL/min.

Exclusion Criteria:

1. Prior systemic therapy or radiation therapy for treatment of the current lung cancer.
2. Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug.
3. Pregnant or lactating female.
4. Unwillingness or inability to follow the procedures required in the protocol.
5. Patients with pre-existing sensorineural hearing impairment/loss or newly diagnosed as documented by an audiology assessment performed prior to study enrollment may not be eligible for cisplatin and may be dispositioned to carboplatin, as determined by the treating physician.
6. Patients with a history of severe hypersensitivity reaction to taxotere and or polysorbate 80 must be excluded.
7. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
8. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
9. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
10. Prior treatment with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody.
11. Known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid indicating acute or chronic infection.
12. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome.
13. History of severe hypersensitivity reaction to any monoclonal antibody and/or to study drug components.
14. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
15. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule.
16. Allergic to contrast agent.
17. Any agents which could affect the absorption or pharmacokinetics of the study drugs.
18. Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate for the study groups | Six months
  Pathologic complete response (pCR) is defined as after neoadjuvant therapy, the surgical specimen can not find any residual cancer cells.
mPR rate for the study groups | Six months
  Major pathologic response (MPR) is defined as pathological less than 10% survival cancer cells after tumor resection.

SECONDARY OUTCOMES:
Toxicity of the study groups | Six months
  Toxicity is assessed by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.
Response rates to neoadjuvant treatment | Six years
  Recurrence-free survival is measured as routine.
Overall survival | Six years
  To correlate major pathologic response with recurrence-free and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China